CLINICAL TRIAL: NCT01551017
Title: Postoperative Cryotherapy: Fast Track Recovery Knee Arthroplasty Project
Brief Title: Fast Track Recovery Knee Arthroplasty Project
Acronym: FARP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: FARP24-214
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Swelling
Keywords: total knee endoprostheses; swelling; mobilisation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- c-treatment: test group
- standard cooling: comparison group

SUMMARY:
Fast Track Recovery Arthroplasty Project is supposed to analyse a new medical method to accelerate patient's remobilisation process after total knee endoprostheses. The method, called c-treatment, is a computer-controlled cryotherapy (soothing cooling therapy) at which the device measures temperature at the affected site (the operated knee in the investigators investigation) and optimizes the cooling temperature. The optimized cooling therapy is supposed to reduce swelling and postoperative pain whereby patient's postoperative mobilization can be done earlier leading to a reduction of length of hospitalization.

To verify c-treatment's efficiency compared to conventional cryotherapy, patients are split in a test group and a standard group. The standard group is treated following the standard protocol at the Department of Orthopaedics Surgery Graz using cold packs (Fa. Dahlhausen, product code 93.000.00.042). Patient's in the test group receive c-treatment therapy following the study protocol.

All patients are instructed to fill in standardized questionnaires to evaluate social scores and pain scores preoperative as well as postoperative. The knee's swelling and range of motion as well as blood parameters monitoring the healing process are measured following the study protocol.

The comparison of these parameters between the standard and the test group is supposed to verify c-treatment's efficiency.

DETAILED DESCRIPTION:
OBJECTIVES

The purpose of this prospective, randomized, single-blind, comparative and controlled clinical study was to evaluate a new cryotherapy device, the cTreatment® system (Waegener®, Belgium) consisting of the Cryoceutical Treatment Server 100 series (CTS) and the Cryoceutical Treatment Pad (cPad®), in comparison to the standard cooling protocol, which was the cold packs (cold/hot pack, Dahlhausen®) currently used at the Department of Orthopaedic Surgery of the Medical University of Graz, Austria, in patients undergoing primary and unilateral TKA surgery. It was particularly focused on the device's efficiency in terms of eventual improvements in the patient's postoperative rehabilitation and mobilisation, such as positive alterations of knee ROM and NRS pain scale, which were set as primary objectives. Further contributing elements, such as alterations of the analgesic consumption, knee girth and the device's safety were set as secondary objectives.

METHODS

Subjects between 18 and 90 suffering from severe degeneratively or traumatically caused gonarthritis or gonarthrosis of the knee joint scheduled for endoprothetic treatment with TKA could be included when giving their informed consent. Exclusion criteria particularly included, on the one side, reasons, which might interfere with the patients' statistical comparability regarding the outcome, such as severe pre-existing local and systemic conditions others than gonarthritis and foregone surgical interventions others than arthroscopy. On the other side it contained conditions, which would interfere with the planned study design, for instance, the standardized medication and PCA and long cooling intervals during hospitalisation.

After giving their written consent they were further randomized to the cryotherapy group, receiving the cTreatment®, or the standard group, receiving cold pack application. Therefore a web-based programme, the "Randomizer", was used (23), considering the patient's sex and scheduled design type of endoprostheses to be implanted, which was either the PFC® or the LCS® (both from DePuy®, Warsaw, IN, USA) endoprosthesis.

After being randomized to the therapy group patients were assigned to the locally applied cryotherapy treatment by use of the cTreatment® system until the end of the clinical study, which was set for POD six. That implied the first cooling session to the extent of one hour already preoperatively on the first preoperative day (PreOD), which coincidently was the day of admission throughout all cases. Furthermore, the subjects received cryotherapy immediately after TKA in the postanaesthesia care unit for six hours in total. During the in-patient setting until POD six the cTreatment® was applied each day for four hours in total, divided into two hours in the morning and two hours in the afternoon. Also there was the option to use the cTreatment® in terms of additional analgesia in the evening for up to four hours on each POD.

PreOD 1 TKA POD 1 POD 2 POD 3 POD 4 POD 5 POD 6

* 1 h pre-OP 6 h post-OP

  4 h optional 2 h morning

  2 h afternoon

  4 h optional 2 h morning

  2 h afternoon

  4 h optional 2 h morning

  2 h afternoon

  4 h optional 2 h morning

  2 h afternoon

  4 h optional 2 h morning

  2 h afternoon

  4 h optional 2 h morning

  2 h afternoon

  4 h optional Table 1: cTreatment® protocol in therapy group

According to the manufacturer, the CTS is a class IIa medical device, which thermodynamically exchanges heat controlled by a built-in computer. It is able to regulate both the flow rate and the fluid's temperature reaching the cPad®. The CTS is operated by use of a touch screen, which allows to start, pause, resume and stop a cooling session. According to the instruction manual the cPad®, which is connected to the Server with flexible tubes using anti-reflux design, is made of flexible Polyurethane, latex free and hypoallergenic. Using hook and loop fasteners it is easy to wrap around the knee ensuring a maximum of contact surface.

The control group was treated abiding by the standard cryotherapy regimen at the Department of Orthopaedic Surgery including the usage of common cold packs (cold/hot pack, Dahlhausen®). They did not receive any cryotherapy before the surgical intervention corresponding to the standard regimen. After TKA cold packs were applied three times per day for 20 minutes each throughout the whole trial. In the context of blinding, the cold packs were placed beneath the applied cPads® in subjects randomized to the standard group, in order to account for a subjectively experienced cold as the CTS was turned off. Besides that, the study setting was identical in both groups.

For the purpose of a better comparability all participating patients received general anaesthesia and a postoperative analgetic therapy based on patient controlled analgesia (PCA), which was filled with diluted hydromorphone, accounting for 0,2 mg hydromorphone per single dose. In addition to that, exclusively Novalgin® 4 x 1 g was administered as a non-opiate analgesic. The PCA was removed after 72 hours postoperative.

The performed physical measurements consisted of the quantification of the knee girth and the ROM of the treated knee joint. The measurements concerning the knee girth were performed at three different levels, at middle-patella, 7 centimetres proximal of the patellar base and 7 centimetres distal of the apex patellae. The ROM was evaluated by use of a hand-held goniometer and the patient being in a supine position. Among the non-physical evaluations was verbally assessing the subjectively experienced pain intensity by use of the eleven-point numeric rating scale (NRS) pain score, about which each patients was told that zero was equal to "no pain at all" and ten was equal to "strongest pain imaginable". The NRS was always evaluated for the state of absolute rest and the state of motion. In this relation the more objectively evaluable analgesics consumption was recorded. Therefore the total hydromorphone usage administered by use of PCA after 72 hours was noted. The physical examinations of the knee joint's ROM and girth and the NRS score evaluation were performed on admission day and POD two, four and six. In the course of the regular change of dressings during the medical rounds the surgical area was exactly examined for potential cold-induced local alterations. In this context, it was particularly searched for signs of frostbite, nerve palsy, inhibited wound healing, deep vein thrombosis and infection. In case of occurrence, the patients had also been told to immediately call attention to eventual adverse effects related to the cold therapy, which they were preliminarily informed about.

IBM® SPSS® Statistics software version 20 was used in order to perform all statistical analyses. In this regard descriptive statistics were conducted using basic calculations of means, standard deviations, ranges, minima and maxima. For the comparisons between the two study groups on admission day, POD two, four and six measured data was first checked for the existence of normal distribution by use of Shapiro-Wilk and Kolmogorov- Smirnov tests. In case of normal distribution, the independent-samples t-test as parametric test was performed. If a normal distribution did not exist, the Wilcoxon-Mann-Whitney test as non-parametric test was performed in order to obtain values of significance regarding between-group distinctions. Throughout the statistical analyses, the level of significance, respectively the P-value was defined as ≤ 0,05.

ELIGIBILITY:
Inclusion Criteria:

* degenerative or posttraumatic gonarthrosis or osteonecrosis around the knee
* scheduled operation for total knee endoprosthesis
* age between 18 and 90 years
* patient agrees with study design, therapy and postoperative controls
* education form is signed by patient and physician

Exclusion Criteria:

* Body Mass Index greater than 40
* varus or valgus deformity greater than 10 degrees
* impaired extension greater than 10 degrees
* flexion preoperative less than 90 degrees
* cold urticaria
* cryoglobulinemia
* paroxysmal cold hemoglobinuria
* current fracture around the knee
* current infection or status post infection
* rheumatoid arthritis at knee
* tumor around the knee
* any operations done around the knee except arthroscopic knee surgery
* active systemic infection (HIV, HBV, HCV)
* obstructive sleep apnea
* opioid intolerance
* incompliance concerning patient controlled analgesia
* cold allergy or cold intolerance
* Raynaud's Disease
* circulatory disorder at the affected leg
* fibromyalgia or other chronic pain syndromes
* taking of immune modulating medication as cortisone, interferon or similar
* depression or anxiety disorder
* addicted to drugs or alcohol
* pregnancy or possible pregnancy without adequate contraception
* no signed education form
* unsoundness of mind

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a total knee endoprosthesis at the Department of Orthopaedics Surgery Graz
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
swelling | preoperative, 2, 4 and 6 days postoperative
  Change in swelling
  swelling is measured ad the midpatellar line as well as seven centimeters distal and seven centimeters proximal of the midpatellar line.
  swelling is measured in centimeters using a standardised measuring tape

SECONDARY OUTCOMES:
Range of motion | preoperative, 2,4 and 6 days postoperative
  Change in Range of motion
  Range of motion is measured with a goniometer using the Neutral position method and compared to previous measured values.
Pain | preoperative, 2,4 and 6 days postoperative
  Change in pain
  pain is evaluated using the Visual Analogue Scale (VAS). The evaluated pain scores are compared to previous pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Glehr, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Orthopaedics Surgery Graz - Medical University Graz, Graz, Austria

REFERENCES:
- [Background] Herbold JA, Bonistall K, Walsh MB. Rehabilitation following total knee replacement, total hip replacement, and hip fracture: a case-controlled comparison. J Geriatr Phys Ther. 2011 Oct-Dec;34(4):155-60. doi: 10.1519/JPT.0b013e318216db81. PMID 22124414
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Sultan PG, Most E, Schule S, Li G, Rubash HE. Optimizing flexion after total knee arthroplasty: advances in prosthetic design. Clin Orthop Relat Res. 2003 Nov;(416):167-73. doi: 10.1097/01.blo.0000081937.75404.ee. PMID 14646757
- [Background] Markert SE. The use of cryotherapy after a total knee replacement: a literature review. Orthop Nurs. 2011 Jan-Feb;30(1):29-36. doi: 10.1097/NOR.0b013e318205749a. PMID 21278552
- [Background] Adie S, Naylor JM, Harris IA. Cryotherapy after total knee arthroplasty a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2010 Aug;25(5):709-15. doi: 10.1016/j.arth.2009.07.010. Epub 2009 Sep 2. PMID 19729279
- [Background] Holmstrom A, Hardin BC. Cryo/Cuff compared to epidural anesthesia after knee unicompartmental arthroplasty: a prospective, randomized and controlled study of 60 patients with a 6-week follow-up. J Arthroplasty. 2005 Apr;20(3):316-21. doi: 10.1016/j.arth.2004.09.043. PMID 15809948